# Statistical Analysis Plan

| TRIAL FULL TITLE | Optimal chemopreventive regimens to prevent malaria and improve birth outcomes in Uganda |
|---|---|
| ClinicalTrials.gov Identifier: | NCT04336189 |
| VERSION | 1.0 |
| VERSION DATE | 20-November-2023 |
| TRIAL STATISTICIAN | Grant Dorsey, MD, PhD Michelle Roh, PhD MPH |
| TRIAL PRINCIPAL INVESTIGATORS | Grant Dorsey, MD, PhD<br>Moses Kamya, MBChB, MMed, PhD<br>Philip Rosenthal, MD |

## **Table of Contents**

| Tā | able o | of Cont | ents2 |
|---|---|---|---|
| 1 | Al | bbrevia | ations and Definitions4 |
| 2 | In | troduc | tion5 |
| | 2.1 | Pre | face5 |
| | 2.2 | Pur | pose of the analyses5 |
| 3 | St | tudy Ob | ojectives and Endpoints6 |
| | 3.1 | Stud | dy Objectives6 |
| | 3.2 | End | points6 |
| | 3.3 | Gen | neral Study Design and Plan |
| | 3.4 | Equ | ivalence or Non-Inferiority Studies |
| | 3.5 | Incl | usion-Exclusion Criteria and General Study Population8 |
| | 3.6 | Ran | domization and Blinding9 |
| | 3.7 | Stud | dy Variables9 |
| | Tabl | le 2. Scl | hedule of routine assessments and procedures in pregnant women9 |
| | Tabl | e 3. St | udy Case Report Forms10 |
| 4 | Sa | ample S | Size10 |
| 5 | G | eneral | Considerations11 |
| | 5.1 | Tim | ing of Analyses11 |
| | 5.2 | Ana | llysis Populations |
| | 5. | .2.1 | Full Analysis Population11 |
| | 5. | .2.2 | Per Protocol Population |
| | 5.3 | Cov | rariates and Subgroups11 |
| | 5.4 | Mis | sing Data12 |
| | 5.5 | Inte | erim Analyses and Data Monitoring12 |
| | 5. | .5.1 | Purpose of Interim Analyses |
| | 5. | .5.2 | Planned Schedule of Interim Analyses12 |
| | Ta | able 4. | Schedule of interim safety analysis and boundaries to monitor study outcome 12 |
| | 5. | .5.3 | Scope of Adaptations |

| | 5.5. | 4 Stopping Rules | .13 |
|---|---|---|---|
| | 5.5. | 5 Adjustment of Confidence Intervals and p-values | .13 |
| | 5.5. | 6 Interim Analysis for Sample Size Adjustment | .13 |
| | 5.5. | 7 Practical Measures to Minimize Bias | .13 |
| | 5.5. | 8 Documentation of Interim Analyses | .13 |
| | 5.6 | Multi-center Studies | . 13 |
| | 5.7 | Multiple Testing | . 13 |
| 6 | Sun | nmary of Study Data | .14 |
| | 6.1 | Trial Profile | . 14 |
| | Tab | le 5. Trial profile | .14 |
| | 6.2 | Baseline Characteristics | . 15 |
| | Tab | le 6. Baseline characteristics of study participants randomized to IPTp | . 15 |
| | 6.3 | Treatment Adherence | . 15 |
| | Tab | le 7. Measures of treatment adherence | .16 |
| 7 | Effic | cacy Analyses (Objectives 1 and 3) | .17 |
| | 7.1 | Efficacy outcomes | . 17 |
| | Tab | le 8. Primary and secondary outcomes | . 17 |
| | 7.2 | Primary Efficacy Analysis | . 19 |
| | Tab | le 9. Outcomes assessed at the time of delivery | .20 |
| 8 | Safe | ety and Tolerability Analyses (Objective 2) | .22 |
| | 8.1 | Adverse Events | . 22 |
| | 8.2 | Serious Adverse Events | . 22 |
| | 8.3 | Analytical Methods | .23 |
| | Tab | le 11. Measures of safety and tolerability | .23 |
| 9 | Refe | erences | .24 |

## **1** Abbreviations and Definitions

| ACT | Artemisinin-based combination therapy |
|------|----------------------------------------------|
| AE | Adverse Event |
| AL | Artemether-lumefantrine |
| CAB | Community advisory board |
| CBC | CBC Complete blood cell |
| CRF | Case Report Form |
| DP | Dihydroartemisinin-piperaquine |
| DSMB | Data and Safety Monitoring Board |
| IDRC | Infectious Diseases Research Collaboration |
| IPT | Intermittent preventive therapy |
| IPTp | Intermittent preventive therapy in pregnancy |
| IRB | Institutional review board |
| LLIN | Long-lasting insecticide treated net |
| MGH | Masafu General Hospital |
| МОН | Ministry of Health |
| MU | Makerere University |
| NIH | National Institute of Health |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SP | Sulfadoxine-pyrimethamine |
| UCSF | University California San Francisco |
| WHO | WHO World Health Organization |

## 2 Introduction

#### 2.1 Preface

Malaria in pregnancy remains a major challenge in Africa, where approximately 50 million women are at risk for *P. falciparum* infection during pregnancy each year. Among pregnant women living in malaria endemic areas characteristic of much of Africa, symptomatic disease is uncommon, but infection with malaria parasites is associated with maternal anemia and adverse birth outcomes including abortions, stillbirth, preterm birth, low birth weight (LBW), and infant mortality. Thus, malaria in pregnancy causes an estimated 900,000 LBW deliveries and 100,000 infant deaths each year. The World Health Organization (WHO) recommends the use of long-lasting insecticidal nets (LLINs) and intermittent preventive treatment with sulfadoxine-pyrimethamine (IPTp-SP) for the prevention of malaria in pregnancy in endemic areas of Africa. However, there is concern for diminishing efficacy of these interventions due to the spread of vector resistance to the pyrethroid insecticides used in LLINs and parasite resistance to SP. Thus, there is an urgent need for new strategies for the prevention of malaria in pregnancy and improving birth outcomes.

Artemisinin-based combination therapies (ACTs) are now the standard treatment for malaria in Africa. Dihydroartemisin-piperaquine (DP) is a fixed-dose ACT and an attractive alternative to SP for IPTp. DP is highly efficacious and the long half-life of piperaquine provides at least 4 weeks of post-treatment prophylaxis. Three randomized controlled trials from our group and others have shown that, compared to IPTp with SP, IPTp with DP dramatically reduced risks of maternal parasitemia and symptomatic malaria, maternal anemia, and placental malaria. In addition, IPTp with DP was as safe and well tolerated as SP. Surprisingly, despite significant reductions in risks of malaria-specific outcomes afforded by DP in these studies, there were no differences between the SP and DP groups in risks of adverse birth outcomes, including LBW and preterm birth. Indeed, in a recent WHO Malaria Policy Advisory Committee concluded that, although IPTp with DP merits further study, SP should remain the recommended drug for IPTp until there is conclusive evidence that alternative regimens improve birth outcomes. Thus, the standard-of-care remains use of a poorly effective antimalarial to prevent malaria in pregnancy.

#### 2.2 Purpose of the analyses

The key question motivating this proposal is why IPTp with either SP or DP is associated with similar risks of adverse birth outcomes despite the far superior antimalarial activity of DP. The likely explanation is that SP, a broad-spectrum antibiotic, protects against non-malarial causes of LBW and preterm birth.<sup>13</sup> In this regard, several studies reported that increased frequency of doses of IPTp with SP was associated with improved birth outcomes and a lower risk of reproductive tract infections (RTIs), despite widespread SP resistance among malaria parasites.<sup>14,15</sup> Our central hypothesis is that SP improves birth outcomes independent of its antimalarial activity and that IPTp with a combination of SP+DP will offer antimalarial and non-antimalarial benefits, thus providing superior prevention of adverse birth outcomes compared to either drug used alone. To test this hypothesis we will conduct a double-blinded randomized clinical trial in a rural area of Uganda with very high malaria transmission intensity where our group already has an established infrastructure for clinical research.

## 3 Study Objectives and Endpoints

## 3.1 Study Objectives

(ICH E3; 8.)

Objective 1: To compare the risk of adverse birth outcomes among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP. We will conduct a randomized controlled trial in 2757 women to test the hypothesis that pregnant women who receive IPTp with SP+DP will have a lower risk of a composite outcome of LBW, preterm birth, small-for-gestational age, fetal loss or neonatal death compared to those who receive either SP or DP alone.

Objective 2: To compare safety and tolerability of IPTp regimens among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP. We will test the hypothesis that pregnant women who receive IPTp with SP+DP will have non-inferior risks of adverse events and measures of tolerability compared to those who receive either SP or DP alone.

Objective 3: To compare risks of malaria-specific and non-malarial outcomes among pregnant women randomized to receive monthly IPTp with SP vs. DP vs. SP+DP. We will test the hypotheses that a) pregnant women who receive IPTp with DP containing regimens will have a lower risk of maternal and placental malaria but a higher risk of *P. falciparum* markers of DP resistance compared to those who receive SP alone; and b) pregnant women who receive IPTp with SP containing regimens will have a lower risk of RTIs and a higher risk of *P. falciparum* markers of SP resistance compared to those who receive DP alone. Further, we will explore impacts of study drugs on the gut and vaginal microbiomes, as differences are likely to impact upon birth outcomes.

## 3.2 Endpoints

(ICH E9; 2.2.2)

## 3.2.1. Primary Outcomes

The primary outcome for objective 1 will be a composite adverse birth outcome, defined as any of the following: spontaneous abortion, stillbirth, LBW, preterm birth, SGA, or neonatal death.

The primary outcome for objective 2 will be the incidence of any grade 3-4 adverse event (AE) or serious adverse event (SAE).

The primary outcome for objective 3a will be the detection of malaria parasites at delivery.

The primary outcome for objective 3b will be the prevalence of reproductive tract infections (RTIs) during pregnancy.

## 3.2.2. Secondary Outcomes

Secondary outcomes for objective 1 will include individual adverse birth outcomes that make up our composite indicator, birthweight, gestational age at delivery, birthweight-for-gestational age z-score, composite of fetal loss and neonatal mortality, and composite adverse birth outcome among live births.

Secondary outcomes for objective 2 will include the incidence of individual AEs, AEs related to study drugs, measures of tolerability of study drugs, congenital anomalies, and maternal mortality.

Secondary outcomes for objective 3a will include measures of malaria, parasitemia, anemia, and DP drug resistance markers during pregnancy.

Secondary outcomes for objective 3b will be changes in the vaginal/gut microbiota, prevalence of STIs/RTIs at delivery, measures of SP drug resistance, change in maternal nutritional status, and gestational weight gain per week.

Study outcomes and definitions are summarized below in Table 1.

**Table 1. Study outcomes** 

| Aim | Outcomes | Definition |
|---|---|---|
| 1 | Composite adverse birth outcome | Spontaneous abortion, stillbirth, LBW, preterm birth, SGA, or neonatal death |
| 1 | Spontaneous abortion | Fetal loss at < 28 weeks gestational age |
| 1 | Stillbirth | Infant born deceased at ≥ 28 weeks gestational age |
| 1 | LBW | Live birth with birth weight < 2500 gm |
| 1 | Preterm birth | Live birth at < 37 weeks gestational age |
| 1 | SGA | Live birth with weight-for-gestational age < 10 <sup>th</sup> percentile of reference population <sup>16</sup> |
| 1 | Neonatal death | Live birth with neonatal death within the first 28 days of life |
| 1 | Birthweight | Birthweight in grams among live births |
| 1 | Gestational age at delivery | Gestational age in weeks estimated by ultrasound among live births |
| 1 | Birthweight-for-gestational age z-score | Birthweight-for-gestational age z-scores among live births. Z-scores calculated based on INTERGROWTH-21st standards <sup>17</sup> |
| 1 | Composite of fetal loss and neonatal mortality | Spontaneous abortion, stillbirth, or neonatal death |
| 2 | Incidence of any grade 3-4 AE or SAE | |
| 2 | Incidence of individual AEs | Based on a standardized AE grading scale <sup>18</sup> |
| 2 | Incidence of AEs related to study drugs | _ |
| 2 | Congenital anomalies | Physical abnormality of live newborn or stillbirths detected at delivery |
| 2 | Maternal mortality | Maternal death up to 4 weeks after delivery |
| 2 | Tolerability of study drugs | Vomiting following administration of study drugs and measures of non-adherence |
| 3a<br> | Detection of malaria parasites at delivery | Parasites detected by microscopy or qPCR in maternal blood, placental blood/tissue |
| 3a | Placental malaria | Detection of malaria parasites or pigment by placental histopathology |
| 3a | Incidence of symptomatic malaria during pregnancy | New episodes of fever plus positive blood smear per person time |
| 3a | Prevalence of parasitemia during pregnancy | Proportion of routine samples with asexual parasites detected by microscopy or qPCR |
| 3a | Prevalence of congenital malaria infection | Proportion of women with parasites detected by microscopy or qPCR in fetal cord blood |
| 3a | Prevalence of anemia during pregnancy | Proportion of routine hemoglobin measurements < 11 g/dL |
| 3a | Prevalence of markers of DP resistance | Proportion of parasite positive samples with molecular markers of DP resistance |
| 3b | Prevalence of STIs/RTIs at delivery | Proportion of vaginal samples collected at delivery positive for STIs/RTIs |
| 3b | Prevalence of markers of SP resistance | Proportion of parasite positive samples with molecular markers of SP resistance |
| 3b | Changes in the vaginal/intestinal microbiota | Relative proportions of different taxonomic groups in vaginal or gut microbiota |
| 3b | Maternal mid-upper arm circumference at last clinic visit before delivery | Mid-upper arm circumference (MUAC) measured at last clinic visit before delivery (continuous; cm); adjusted for values measured on the day study drugs first given |
| 3b | Gestational weight gain per week | Maternal weight measured at the last clinic visit before delivery minus the maternal weight at on the day study drugs first given, divided by the number of weeks between those dates; adjusted for values on the day study drugs first given |

## Study methods

## 3.3 General Study Design and Plan

(ICH E3;9)

This will be a double-blinded randomized controlled phase III trial of 2757 HIV uninfected pregnant women. HIV uninfected women at 12-20 weeks gestation will be randomized in equal proportions to one of three IPTp treatment arms: 1) SP given every 4 weeks, or 2) DP given every 4 weeks, or 3) SP+DP given every 4 weeks. SP or DP placebos will be used to ensure adequate blinding is achieved. Follow-up for the pregnant women will end 28 days after giving birth.

Recruitment will take place in two phases. In phase 1, 300 participants will be enrolled over 2-3 months. Phase 1 participants will undergo intensive safety and pharmacokinetic assessment. At the end of phase 1, an interim analysis of safety data will be performed and presented to the Data and Safety Monitoring Board (DSMB) as described in detail in the Protection of Human Subjects section and study protocol. If the DSMB approves, phase 2 of recruitment will begin and continue until the target sample size has been reached.

## 3.4 Equivalence or Non-Inferiority Studies

(ICH E3; 9.2, 9.7.1, 11.4.2.7. ICH E9; 3.3.2)

N/A - This trial is designed as a superiority trial.

## 3.5 Inclusion-Exclusion Criteria and General Study Population

(ICH E3;9.3. ICH E9;2.2.1)

## 3.5.1. Inclusion Criteria

- 1) Viable singleton pregnancy confirmed by ultrasound
- 2) Estimated gestational age between 12-20 weeks
- 3) Confirmed to be HIV uninfected by rapid test
- 4) 16 years of age or older
- 5) Resident of Busia District, Uganda
- 6) Provision of informed consent
- 7) Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
- 8) Willing to deliver in the hospital

#### 3.5.2. Exclusion Criteria

- 1) History of serious adverse event to SP or DP
- 2) Active medical problem requiring inpatient evaluation at the time of screening
- 3) Intention of moving outside of Busia District, Uganda
- 4) Chronic medical condition requiring frequent medical attention
- 5) Prior chemopreventive therapy or any other antimalarial therapy during this pregnancy
- 6) Early or active labor
- 7) Multiple pregnancies (i.e. twins/triplets)

## 3.6 Randomization and Blinding

(ICH E3; 9.4.3, 9.4.6. ICH E9; 2.3.1, 2.3.2)

There will be 3 treatment arms for the woman during pregnancy; SP given every 4 weeks, DP given every 4 weeks or a combination of SP+DP given every 4 weeks. We will use a 1:1:1 randomization scheme targeting 919 pregnant women in each treatment arm. A randomization list will be computer generated by a member of the project who will not be directly involved in the conduct of the study. The randomization list will include consecutive treatment numbers with corresponding random treatment assignments. Randomized codes will correspond to the 3 treatment arms using permuted variable sized blocks of 6 and 9. Sealed copies of the original randomization list and documentation of the procedure used to generate the lists will be stored in the project administrative offices in San Francisco and Kampala. Prior to the onset of the study, a set of sequentially numbered, opaque, sealed envelopes will be prepared. Each envelope will be marked on the outside with the treatment allocation number. The inside of the envelope will contain a piece of paper with the treatment allocation number and treatment group assignment along with a piece of carbon paper.

## 3.7 Study Variables

(ICH E3; 9.5.1. ICH E9; 2.2.2)

Table 2. Schedule of routine assessments and procedures in pregnant women

| Evaluations and Interventions | Enrollment | | | ٧ | Veeks c | of gestat | ion | | | Delivery | 1 and 4 weeks |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Evaluations and interventions | Enrollment | 16* | 20 | 24 | 28 | 29 | 32 | 36 | 40 | Delivery | postpartum |
| Informed consent | Х | | | | | | | | | | |
| HIV testing <sup>1</sup> | Х | | | | | | | | | Х | |
| Obstetrical ultrasound <sup>2</sup> | Х | | | Х | | | Х | X** | | | |
| Blood collected by phlebotomy for CBC | Х | | Х | | Х | | | Х | | Х | |
| Blood collected by finger prick for blood | Х | Х | Х | Х | Х | | Х | Х | х | Х | |
| smear and dried blood spot | | | | | | | | | | | |
| Routine assessment in the study clinic <sup>3</sup> | Х | Х | Χ | Х | Χ | | Х | Х | Х | | X |
| ECG testing and collection of plasma samples | | | x | | x | | | x | | | |
| for PK studies (phase 1 only)4 | | | , | | , | | | , | | | |
| Administration of study drugs | | Х | Х | Χ | Х | | Х | Х | Х | | |
| Collection of cord blood and placental | | | | | | | | | | x | |
| blood/tissue | | | | | | | | | | ^ | |
| Labor and delivery documentation <sup>5</sup> | | | | | | | | | | Х | |
| Collection of gut and vaginal samples for | Х | | | | | X** | Х | | | | |
| microbiome studies | ^ | | | | | _ ^ | _ ^ | | | | |
| Collection samples for testing of STIs/RTIs | | | | | | | | | | Х | |
| Standard Care | | | | | | | | | | | |
| Obstetrical exam <sup>6</sup> | Х | Х | Х | Х | Х | | Х | Х | Х | Х | Х |
| Syphilis screening | Х | | | | | | | | | | |
| Iron and Folic Acid | Х | Х | Х | Χ | Х | | Х | Х | Х | | |
| Prenatal vitamins | Х | | | | | | | | | | |
| Mebendazole <sup>7</sup> | | Х | | | | | | | | | |
| Vitamin A <sup>8</sup> | | | | | | | | | | Х | |
| Insecticide treated bednet | Х | | | | | | | | | | |

<sup>\*</sup> Only if study subject enrolled prior to 16 weeks gestation

<sup>\*\*</sup> For a subset of individuals

#### **Explanation of maternal schedule of events**

- 1. HIV test will be done at enrollment and documented. A repeat rapid HIV test will be done at delivery. HIV testing shall be done using standard rapid HIV-testing algorithm.
- 2. Ultrasound will be done to confirm intrauterine pregnancy and estimate gestational age at enrollment.
- 3. Targeted physical exam will include anthropometric measurements (e.g. weight) and vital signs (i.e. temperature, pulse, and blood pressure). Measurement of height at the enrollment visit only.
- 4. For women enrolled in phase 1 of the study, pre- and post-study drug ECG will be performed and finger-prick blood samples will be collected to measure piperaquine levels.
- 5. Labor & Delivery documentation will include: Peripartum history, mode of delivery, Apgar scores (when available), weight, length, and head circumference of the child at birth, approximate gestational age, duration of labor, signs of fetal distress (presence of meconium), summary of events in first days of life (including feeding, breathing patterns, jaundice, lethargy, or any additional abnormal findings), duration of admission if delivered in hospital.
- 6. Obstetrical exam includes estimation of gestational age at study entry, fundal height measurement, fetal heart tones and urine dipstick for protein. A cervical exam will also be performed at screening and during antepartum study visits as clinically indicated.
- 7. Mebendazole is typically given as 500mg as a single dose as early as possible after the 1<sup>st</sup> trimester (16 or 20 week visit).
- 8. Vitamin A supplementation is dosed as 200,000 IU.

**Table 3. Study Case Report Forms** 

| Screening Form |
|---------------------------------------------|
| Enrollment Form |
| Clinic Visit Form |
| AE Form |
| Mother Delivery Form |
| Ultrasound Form |
| Placental Histopathology Form |
| Hospital Admission Form |
| Postpartum Form |
| Study Drug Dispensing Form |
| Subject Death Form |
| Subject Withdrawal or Study Completion Form |
| ECG Form |

## 4 Sample Size

(ICH E3; 9.7.2. ICH E9; 3.5)

Our sample size calculation is based on testing the primary hypothesis for specific aim 1. Based on our previous study from the same site, the risk of the composite adverse birth outcome as defined for aim 1 was 22.6% in the SP and 25.1% in the DP arm among women meeting the eligibility criteria Statistical Analysis Plan version 1.0: Optimizing IPTp in Uganda


for this proposal. Given these estimates, we would need to enroll 2757 women (assuming 15% loss to follow-up) to have 80% power (2-sided alpha = 0.05) to detect a 25% or greater reduction in the risk of our composite adverse birth outcome in the SP+DP arm compared to either of the other arms. For the primary outcome of specific aim 2, we assume that the incidence of any grade 3-4 AE or SAE will be 0.37 per person year (SD=0.57) in the SP arm and 0.18 per person year (SD=0.35) in the DP arm, based on our previous study. Given these estimates we will have 80% power (1-sided alpha = 0.025) for our non-inferiority margin to be set at 0.07 when comparing the SP+DP arm to the SP arm and at 0.03 when comparing the SP+DP arm to the DP arm. For the primary outcome of specific aim 3a, we assume that the risk of detection of malaria parasites at delivery will be 12.5% in the SP arm based on our previous study. Given our sample size, we will have 80% power (2-sided alpha = 0.05) to detect a 32% or greater reduction in the prevalence of malaria parasites at delivery in the SP+DP arm or the DP arm compared to the SP arm.

## 5 General Considerations

## 5.1 Timing of Analyses

The final trial analysis for the study will be performed after the last enrolled woman has given birth, complete 4 weeks of follow-up postpartum, and all outcome measures have been assessed. Prior to the final analysis we will perform an interim safety analysis when the first 300 women enrolled have been followed through delivery (phase 1) and then every 6 months during phase 2 of the study. The interim safety analyses will compare the incidence of significant adverse events (grade 3/4 & SAEs).

## **5.2** Analysis Populations

(ICH E3; 9.7.1, 11.4.2.5. ICH E9; 5.2)

A modified intention-to-treat approach to all analyses will be used, including all study participants randomized to therapy and have the outcome of interest measured including all follow-up time until the study participant completes the study or early study termination regardless of whether the intervention was stopped due to an adverse event. Analyses for safety and tolerability endpoints will be conducted using a subset of the modified intention-to-treat population, consisting of all randomised subjects who received at least one dose of the study drug. All subjects will be analysed according to their randomized treatment arm.

#### 5.2.1 Full Analysis Population

- All subjects who were randomized
- All subjects with evaluable data on specific outcomes

#### 5.2.2 Per Protocol Population

A per protocol analysis is not planned.

#### 5.3 Covariates and Subgroups

(ICH E3; 9.7.1, 11.4.2.1. ICH E9; 5.7)

Covariates of interest will include baseline measures of maternal age, gestational age at enrollment, gravidity, LLIN ownership, socio-economic status as estimated by a household wealth index, and prevalence of malaria parasites.

Sub-group analyses will be performed based on categories of maternal age, gravidity, infant sex, and gestational age at the time study drugs were first administered.

## 5.4 Missing Data

(ICH E3; 9.7.1, 11.4.2.2. ICH E9;5.3. EMA Guideline on Missing Data in Confirmatory Clinical Trials)

Women in the trial who are prematurely withdrawn from the study or are not able to provide data for specific outcomes will be considered un-evaluable and will not be included in the primary trial analysis.

## 5.5 Interim Analyses and Data Monitoring

(ICH E3; 9.7.1, 11.4.2.3. ICH E9; 4.1, FDA Feb 2010 "Guidance for Industry Adaptive Design Clinical Trials for Drugs and Biologics")

## **5.5.1** Purpose of Interim Analyses

Over the course of the trial, we will perform interim safety analyses when the first 300 women enrolled have been followed through delivery (phase 1) and then every 6 months during phase 2 of the study. The interim safety analyses will compare the incidence rate ratio of significant adverse events (grade 3/4 & SAEs). The interim analyses will not include an evaluation of efficacy outcomes.

## **5.5.2** Planned Schedule of Interim Analyses

An interim safety analysis for pregnant women will be performed when the first 300 women enrolled have been followed through delivery (phase 1) and then every 6 months during phase 2 of the study. A standardized test statistic will be calculated for the incident rate ratio of significant adverse events (grade 3/4 & SAEs). If this statistic exceeds the nominal critical value calculated using the error spending function (Table 4), then a statistically significant result will have been achieved at the time of the analysis. In that event, the sponsor will be notified and a report submitted for review by the Data Safety Monitoring Board (DSMB). For the interim safety analyses, the study team will present information on recruitment and the results of interim safety analyses to the DSMB, which will review the data and recommend a course of action.

Table 4. Schedule of interim safety analysis and boundaries to monitor study outcome

| Number of Evaluable Subjects Accrued | Test Sta | tistic | Alpha | Cumulative |
|---|---|---|---|---|
| Number of Evaluable Subjects Actifued | Lower Bound | <b>Upper Bound</b> | Aipiia | Alpha |
| N=300 (phase 1) | -5.37 | 5.37 | 0.000001 | 0.0000001 |
| N=791 (phase 2) | -3.71 | 3.71 | 0.0002069 | 0.000207 |
| N=1282 (phase 2) | -2.97 | 2.97 | 0.002844 | 0.003051 |
| N=1773 (phase 2) | -2.54 | 2.54 | 0.009046 | 0.0121 |
| N=2264 (phase 2) | -2.25 | 2.25 | 0.01605 | 0.02815 |
| N=2757 or 100% of accrual | -2.04 | 2.04 | 0.02185 | 0.05 |

This analysis assumes  $\alpha$ =0.05 (two-sided test), O'Brien-Fleming boundaries (DeMets error-spending function) and 2757 trial participants. We will utilize Programs for Computing Group Sequential Boundaries Using the Lan-DeMets Method.

#### 5.5.3 Scope of Adaptations

At the time of the interim analyses, the DSMB may decide to continue, stop, or modify the trial based on the interim safety analysis. This may include the discontinuation of a study arm and rerandomization or cessation of subject participation in the stopped arm.

#### 5.5.4 Stopping Rules

The DSMB will determine whether to stop the study for early evidence of intervention safety problems after a thorough review of interim data. Interim reports will provide cumulative enrollment figures and cumulative adverse birth outcomes, serious adverse events (classified according to grade), sorted by study arm. Brief clinical descriptions of key events will also be provided. The PIs will be responsible for immediately reporting to the funding agency any temporary or permanent suspension of the project and the reason for the suspension.

#### 5.5.5 Adjustment of Confidence Intervals and p-values

As appropriate we will adjust p-values and confidence intervals taking into account the specified error spending functions and interim evaluation of the data.

#### 5.5.6 Interim Analysis for Sample Size Adjustment

The sample size will not be adjusted based on the results of the interim analysis.

#### 5.5.7 Practical Measures to Minimize Bias

The study will establish and control who will have access to what information at each stage of the trial. Uncontrolled reporting of interim analyses to study investigators responsible for recruiting subjects will not occur.

The following measure will be taken to minimize bias:

- Only the study statistician and assistant statistician will perform the interim analysis.
- Only the statisticians and the DSMB will see any data or analyses at the interim analysis
- No information will be publicly available following an interim analysis
- Information will be provided to the sponsor and investigators as per recommendation of the study DSMB.
- Only the statisticians will be unblinded at for the interim analysis

## **5.5.8** Documentation of Interim Analyses

Snapshots of the data available at each interim analysis will be preserved, as will all documentation of analysis plans, programming code and reporting provided at the interim analysis.

## 5.6 Multi-center Studies

(ICH E3;9.7.1, 11.4.2.4. ICH E9; 3.2)

This is a single center study.

## 5.7 Multiple Testing

(ICH E3; 9.7.1, 11.4.2.5. ICH E9; 2.2.5)

This study has one primary outcome for each objective and multiple secondary outcomes. No formal adjustment of p-values and confidence intervals will be made for the comparison of multiple a priori outcomes.

## 6 Summary of Study Data

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, interquartile range, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. All summary tables will be structured with a column for each treatment and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

#### **6.1** Trial Profile

The overall study profile will be presented as a figure following CONSORT guidelines. The total numbers of women screened, excluded during screening (including criteria for exclusion) and enrolled will be presented. The numbers of women enrolled in each treatment arm and followed through each stage of the trial profile are presented in skeleton Table 5 below.

**Table 5. Trial profile** 

| Screened | | ### | |
|-------------------------------------------|-----|---------------|-------|
| Excluded during screening* | | ### | |
| | | Treatment arm | |
| | SP | DP | DP+SP |
| Enrolled and randomized | ### | ### | ### |
| Withdrawn before receiving study drugs* | ### | ### | ### |
| Received at least one dose of study drugs | ### | ### | ### |
| Withdrawn before delivery* | ### | ### | ### |
| Delivered | ### | ### | ### |
| Withdrawn after delivery* | ### | ### | ### |
| Completed 4-week post-partum visit | ### | ### | ### |

<sup>\*</sup> Specific reasons for exclusion or withdrawal will be reported

#### **6.2** Baseline Characteristics

Skeleton table of all baseline variables collected on the day of enrollment that will be presented are provided in Table 6 below.

Table 6. Baseline characteristics of study participants randomized to IPTp

| | Treatment arm | | |
|---|---|---|---|
| Characteristic | SP | DP | DP+SP |
| | (n=XXX) | (n=XXX) | (n=XXX) |
| Age in years, mean (SD) | | | |
| Gestational age in weeks, mean (SD) | | | |
| Gestational age categories, n (%) | | | |
| 12-16 weeks | | | |
| >16-20 weeks | | | |
| Gravidity, n (%) | | | |
| 1 | | | |
| 2 | | | |
| <u>≥</u> 3 | | | |
| Bednet ownership, n (%) | | | |
| None | | | |
| Untreated net | | | |
| Long-lasting insecticide-treated net | | | |
| Household wealth index, n (%) | | | |
| Lowest tertile | | | |
| Middle tertile | | | |
| Highest tertile | | | |
| Weight in kg, mean (SD) | | | |
| Height in cm, mean (SD) | | | |
| Maternal MUAC, mean (SD) | | | |
| Maternal malnutrition, n (%) | | | |
| Laboratory values, mean (SD) | | | |
| WBC count per mm <sup>3</sup> | | | |
| Neutrophil count per mm <sup>3</sup> | | | |
| Platelet count per mm <sup>3</sup> | | | |
| Hemoglobin g/dL | | | |
| Detection of malaria parasites by microscopy, n (%) | | | |
| Detection of malaria parasites by microscopy or qPCR, n (%) | | | |

#### **6.3** Treatment Adherence

During pregnancy, women will be given 1 of 3 treatment regimens: 1) SP given every 4 weeks during pregnancy, 2) DP given every 4 weeks, or 3) SP+DP given every 4 weeks during pregnancy. Each treatment with SP will be given as a single dose consisting of 3 full strength tablets. Each treatment with DP will consist of 3 full strength tablets given once a day for 3 consecutive days. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo, DP and placebo, or SP and DP) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP. Administration of all study drugs will be double blinded such that study participants and study staff will be blinded to study treatments with the exception of the study pharmacist and pharmacy technician, who will not be involved with patient care or assessment Statistical Analysis Plan version 1.0: Optimizing IPTp in Uganda


of study outcomes. All doses of study drugs will be pre-packaged by a study pharmacist and administered by a study nurse blinded to the study participant's treatment regimen. All doses of SP (or SP placebo) administered will be directly observed in the clinic. For DP (or DP placebo), the first of the 3 daily doses will be directly observed in the clinic and the 2<sup>nd</sup> and 3<sup>rd</sup> daily doses will be administered at home using pre-packaged study drugs in opaque envelopes with dosing instructions written on the outside. For doses of study drugs administered in the clinic, if a study participant vomits the study drug within 30 minutes of administration, the drug will be re-administered. For doses of study drugs administered at home, if a study participant vomits the study drug within 30 minutes of administration or study drug is lost, the study participant will be instructed to come to the study clinic as soon as possible where the study drug will be re-administered/replaced. For pregnant women all doses of study drugs will be given between 16 and 40 weeks gestation. Measures of treatment adherence are summarized in skeleton Table 7 below.

Table 7. Measures of treatment adherence and tolerability

| | 7 | Treatment arm | |
|---|---|---|---|
| | SP | DP | DP+SP |
| At the level of each individual woman receiving at least one of | dose of study o | drugs | |
| At least one dose of study drug held for adverse event | n/N (%) | n/N (%) | n/N (%) |
| Missed at least 1 course of study drugs (all 3 doses) | n/N (%) | n/N (%) | n/N (%) |
| Reported not taking at least 1 dose of study drug at home | n/N (%) | n/N (%) | n/N (%) |
| At least one dose of study drug vomited | n/N (%) | n/N (%) | n/N (%) |
| At the level of each scheduled dose of study of | lrug | | |
| Study drugs (all 3 doses) held for adverse event | n/N (%) | n/N (%) | n/N (%) |
| Study drugs (all 3 doses) missed | n/N (%) | n/N (%) | n/N (%) |
| Vomited day 1 dose of study drugs (observed) | n/N (%) | n/N (%) | n/N (%) |
| Reported not taking day 2 dose of study drugs at home | n/N (%) | n/N (%) | n/N (%) |
| Reported vomiting day 2 dose of study drugs at home | n/N (%) | n/N (%) | n/N (%) |
| Reported not taking day 3 dose of study drugs at home | n/N (%) | n/N (%) | n/N (%) |
| Reported vomiting day 3 dose of study drugs at home | n/N (%) | n/N (%) | n/N (%) |

## 7 Efficacy Analyses (Objectives 1 and 3)

## 7.1 Efficacy outcomes

Definitions and criteria used to generate estimates of all primary and secondary efficacy outcomes are presented in Table 8 below.

**Table 8. Primary and secondary outcomes** 

| Outcome | Category | Type of measurement | Timing of measurement | Numerator | Denominator | Missing data |
|---|---|---|---|---|---|---|
| Composite adverse birth outcome | Primary outcome objective 1 | Proportion | At delivery and 28 days postpartum | Any of the following: spontaneous abortion, stillbirth, low birth weight, preterm delivery, small for gestational age, or neonatal death | All women who deliver | Withdrawn prior to delivery |
| Low birth weight | Secondary<br>outcome<br>objective 1 | Proportion | At delivery | Birth weight < 2500 gm | Deliveries with a live birth | Withdrawn prior to delivery or deliveries with fetal loss |
| Preterm delivery | Secondary<br>outcome<br>objective 1 | Proportion | At delivery | Gestational age < 37 weeks | Deliveries with a live birth | Withdrawn prior to delivery or deliveries with fetal loss |
| Small for gestational age | Secondary<br>outcome<br>objective 1 | Proportion | At delivery | < 10 <sup>th</sup> percentile based on INTERGROWTH-<br>21 <sup>st</sup> standards <sup>17</sup> | Deliveries with a live birth | Withdrawn prior to delivery or deliveries with fetal loss |
| Spontaneous abortion | Secondary<br>outcome<br>objective 1 | Proportion | At delivery | Delivery at < 28 weeks gestational age | All deliveries | Withdrawn prior to delivery |
| Stillbirth | Secondary<br>outcome<br>objective 1 | Proportion | At delivery | Infant born deceased | Deliveries ≥ 28 weeks gestational age | Withdrawn prior to delivery or < 28 weeks gestational age |
| Neonatal death | Secondary<br>outcome<br>objective 1 | Proportion | 28 days postpartum | Infant death in the first 28 days of life | Deliveries with a live birth | Withdrawn prior to delivery or deliveries with fetal loss |
| Birthweight | Secondary<br>outcome<br>objective 1 | Mean, quantile | At delivery | Mean birthweight in grams among live births, 650th, and 90th percentile) among live births | ean birthweight in grams among live births, differences in birthweight quantiles (i.e., $10^{\rm th}$ , and $90^{\rm th}$ percentile) among live births | |
| Gestational age at delivery | Secondary<br>outcome<br>objective 1 | Mean | At delivery | Mean gestational age in weeks among live birt | hs | Withdrawn prior to delivery or deliveries with fetal loss |
| Birthweight-for-<br>gestational age Z-score | Secondary<br>outcome<br>objective 1 | Mean | At delivery | Birthweight-for-gestational age z-scores amon<br>INTERGROWTH-21 <sup>st</sup> standards <sup>17</sup> | g live births. Z-scores calculated based on | Withdrawn prior to delivery or deliveries with fetal loss |
| Composite of fetal loss and neonatal mortality | Secondary<br>outcome<br>objective 1 | Proportion | At delivery and 28 days postpartum | Any of the following: spontaneous abortion, stillbirth, or neonatal death | All women who deliver | Withdrawn prior to delivery |

| Detection of malaria parasites at delivery | Primary<br>outcome<br>objective 3a | Proportion | At delivery | Any malaria parasites detected by microscopy or qPCR from maternal blood, placental blood, or placental tissue collected at delivery | Number of deliveries with samples collected | Withdrawn prior to delivery or no delivery samples collected |
|---|---|---|---|---|---|---|
| Detection of placental malaria | Primary<br>outcome<br>objective 3a | Proportion | At delivery | Any evidence of malaria parasites or pigment by placental histopathology | All women who deliver | Withdrawn prior to delivery or failure to collect samples for placental histopathology |
| Incidence of symptomatic malaria during pregnancy | Secondary<br>outcome<br>objective 3a | Incidence | Time at risk during pregnancy | Number of episodes of fever and positive blood smear by microscopy | Duration of observation from day following<br>1st dose of study drugs to delivery or<br>premature study withdrawal | None |
| Prevalence of parasitemia during pregnancy | Secondary<br>outcome<br>objective 3a | Proportion | At the time of each routine visit | Maternal blood samples with parasites detected by microscopy or qPCR | Routine visits at 20, 24, 28, 32, 36, and 40 weeks of gestational age following 1st dose of study drugs to delivery or premature study withdrawal | Missed routine visits or samples not collected |
| Prevalence of congenital malaria infection | Secondary<br>outcome<br>objective 3a | Proportion | At the time of delivery | Presence of parasites detected by microscopy or PCR in fetal cord blood | All women who deliver | Withdrawn prior to delivery, fetal cord blood not collected, |
| Maternal anemia | Secondary<br>outcome<br>objective 3a | Proportion | At the time of each<br>routine visit and at<br>delivery when<br>phlebotomy done | Hemoglobin level < 11 g/dL | Routine visits at 20,28, 36 weeks of gestational age following 1st dose of study drugs to delivery or premature study withdrawal | Missed routine visits or sample not collected when scheduled for phlebotomy |
| Prevalence of molecular<br>markers of DP<br>resistance | Secondary<br>outcome<br>objective 3a | Proportion | At the time of each routine visit or when malaria diagnosed | Detection of malaria parasites containing molecular markers of DP resistance | Detection of malaria parasites following 1st dose of study drugs | Samples where malaria parasites<br>detected but assays for molecular<br>markers of DP resistance failed |
| Prevalence of STIs/RTIs | Primary<br>outcome<br>objective 3b | Proportion | At the time of delivery | Women who deliver and test positive for the presence of STIs/RTIs | Women who deliver and successfully tested for the presence of STIs/RTIs | Failure to collect samples at delivery or failure to generate results |
| Changes in vaginal/gut microbiome | Secondary<br>outcome<br>objective 3b | Abundance of microorganisms | At enrollment and at 36 weeks gestational age | Changes in relative and absolute abundance of | es in relative and absolute abundance of microorganisms | |
| Prevalence of molecular<br>markers of SP<br>resistance | Secondary<br>outcome<br>objective 3b | Proportion | At the time of each routine visit or when malaria diagnosed | Detection of malaria parasites containing molecular markers of SP resistance | Detection of malaria parasites following 1st dose of study drugs | Samples where malaria parasites<br>detected but assays for molecular<br>markers of SP resistance failed |
| Maternal MUAC at last clinic visit before delivery | Secondary<br>outcome<br>objective 3b | Mean | At enrollment and at last clinic visit before delivery | Mid-upper arm circumference (MUAC) values m<br>adjusted for MUAC values on the day study dru<br>until > 27 weeks gestational age (3 <sup>rd</sup> trimester) | Failure to collect MUAC values on the day study drugs first given | |
| Gestational weight gain<br>per week | Secondary<br>outcome<br>objective 3b | Mean | At each clinic visit<br>(from enrollment to<br>delivery) | Maternal weight measured at the last clinic visit<br>the day study drugs first given, divided by the n<br>adjusted for weight on the day study drugs first<br>until > 27 weeks gestational age (3 <sup>rd</sup> trimester) | Failure to collect weight values on the day study drugs first given | |


## 7.2 Primary Efficacy Analysis

#### **Objective 1**

For objective 1, we will test the hypothesis that pregnant women who receive IPTp every 4 weeks with a combination of SP+DP will have a lower risk of our composite adverse birth outcome compared to those who receive either SP or DP alone.

**Primary analysis.** Using a modified intent-to-treat approach, we will compare the prevalence of our primary outcome between the study arms using unadjusted log-binomial models. Results will be presented as the risk ratio (RR) or reduction of the RR (1-RR x 100%) if the RR is lower than 1. We will explore for any differences of potential confounders between the treatment arms and if necessary adjust our analysis using multivariate log-binomial models. If the log-binomial model does not converge, modified Poisson regression with robust standard errors will be used to estimate RR.

**Secondary analyses.** For secondary binary outcomes, we will compare the prevalence of our individual adverse birth and neonatal outcomes using the same approach as our primary analysis. For comparing secondary continuous outcomes, linear regression will be used to compare differences between arms. Quantile regression may also be used if assumptions for linear regression cannot be met (e.g., linearity, homoscedasticity, independence, or normality) and to determine whether treatment arms were associated with nuanced changes in the lower and upper percentiles distribution of continuous outcomes (e.g., changes in the 10<sup>th</sup> or 90<sup>th</sup> percentile of birthweight). For outcomes that that were also measured at enrollment (e.g., fetal weight), enrollment measures will be included as a covariate in the model.

For subgroup analyses, we will include a two-way interaction term between treatment arm and subgroup of interest in our models. If the p-value of the interaction term is less than 0.1, we will consider this finding to be statistically significant. For all other p-values, values less than 0.05 will be considered statistically significant.

#### **Objective 3**

For objective 3a, we will test the hypotheses that pregnant women who receive IPTp regimens containing DP will have a lower risk of measures of malaria during pregnancy and at delivery but a higher risk of infection with malaria parasites containing mutations associated with DP resistance compared to those who receive SP alone. For objective 3b, we will test the hypotheses that pregnant women who receive IPTp regimens containing SP will have a lower risk of STIs/RTIs, greater changes in their vaginal/intestinal microbiota, improved maternal nutrition, and a higher risk of infection with malaria parasites containing mutations associated with SP resistance compared to those who receive DP alone.

**Analysis.** We will compare proportions between the study arms using log-binomial models and presented as the risk ratio (RR) or reduction of the RR (1-RR x 100%) if the RR is lower than 1. For repeated measures in the same study participant (parasite prevalence and anemia during pregnancy,

prevalence of molecular markers of drug resistance) we will use generalized estimating equations with a log-binomial model and robust standard errors. We will compare the incidence of malaria during pregnancy using negative binomial regression models. These models will include the logarithm of the follow-up time as an offset. We will translate the fitted coefficients and their confidence bounds into percentage effects with the formula 100\*[exp(coefficient)-1]. This approach is closely related to exponential survival models for analyzing events per follow-up time, but is better able to adjust for violated assumptions. If necessary, multivariate analyses will be performed to adjust for potential confounders and effect modifiers. The main results will be based on the adjusted analyses if residual confounding is present. Comparisons of incidence measures will be expressed at the incidence rate ratio (IRR) or the protective efficacy (PE = 1-IRR x 100%). For continuous outcomes, either linear regression or quantile regression will be used to compare differences between arms, with a similar rationale to those stated in Objective 1. For outcomes that that were also measured at enrollment (e.g., fetal weight), enrollment measures will be included as a covariate in the model. Subgroup analyses will be conducted using the same approach as Objective 1.

Skeleton tables for the presentation of primary and secondary efficacy outcomes are presented in Tables 9-11 below.

Table 9. Composite primary outcome and its components assessed at the time of delivery

| | Treatment arm | | | | | | |
|---|---|---|---|---|---|---|---|
| Outcome | SP <sup>a</sup> DP | | | | DP+SP | | |
| | Prevalence | Prevalence | RR (95% CI) | p-value | Prevalence | RR (95% CI) | p-value |
| Composite adverse birth outcome | n/N (%) | n/N (%) | | | n/N (%) | | |
| Individual birth outcomes | | | | | | | |
| Spontaneous abortion | n/N (%) | n/N (%) | | | n/N (%) | | |
| Stillbirth | n/N (%) | n/N (%) | | | n/N (%) | | |
| Low birth weight | n/N (%) | n/N (%) | | | n/N (%) | | |
| Preterm delivery | n/N (%) | n/N (%) | | | n/N (%) | | |
| Small for gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| Neonatal death | n/N (%) | n/N (%) | | | n/N (%) | | |
| Fetal or neonatal loss | n/N (%) | n/N (%) | | | n/N (%) | | |

<sup>&</sup>lt;sup>a</sup> Reference group

Table 10. Secondary efficacy outcomes assessed at the time of delivery

| | Treatment arm | | | | | | |
|---|---|---|---|---|---|---|---|
| Outcome | SP <sup>a</sup> DP | | | SP+DP | | | |
| | Mean (SD) | Mean (SD) | MD (95% CI) | p-value | Mean (SD) | MD (95% CI) | p-value |
| Birthweight in grams | XX (XX) | XX (XX) | | | XX (XX) | | |
| Gestational age at delivery in weeks | XX (XX) | XX (XX) | | | XX (XX) | | |
| Birthweight-for-gestational age z-score | XX (XX) | XX (XX) | | | XX (XX) | | |
| Maternal MUAC in cm <sup>b</sup> | XX (XX) | XX (XX) | | | XX (XX) | | |
| | Prevalence | Prevalence | RR (95% CI) | p-value | Prevalence | RR (95% CI) | p-value |
| Detection of malaria parasites at delivery | n/N (%) | n/N (%) | | | n/N (%) | | |
| Detection of placental malaria | n/N (%) | n/N (%) | | | n/N (%) | | |
| Detection of congenital malaria infection | n/N (%) | n/N (%) | | | n/N (%) | | |
| Prevalence of STIs/RTIs at delivery | n/N (%) | n/N (%) | | | n/N (%) | | |
| | | | | | • | | |

<sup>&</sup>lt;sup>a</sup> Reference group

<sup>&</sup>lt;sup>b</sup> Adjusted for baseline values

 Table 11. Longitudinal secondary outcomes assessed during pregnancy

| Outcome | Treatment arm | | | | | | |
|---|---|---|---|---|---|---|---|
| Outcome | SP a DP | | | | SP+DP | | |
| Incidence measures | Events <sup>b</sup> | Events <sup>b</sup> | IRR<br>(95% CI) | p-<br>value | Events <sup>b</sup> | IRR<br>(95% CI) | p-<br>value |
| Symptomatic malaria | xx (x.xx) | xx (x.xx) | | | xx (x.xx) | | |
| Prevalence measures | Prevalence | Prevalence | RR<br>(95% CI) | p-<br>value | Prevalence | RR<br>(95% CI) | p-<br>value |
| Detection of malaria parasites by microscopy or qPCR | | | | | | | |
| All routine visits | n/N (%) | n/N (%) | | | n/N (%) | | |
| 20 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 24 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 28 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 32 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 36 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 40 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| Anemia defined as hemoglobin level < 11 g/dL | | | | | | | |
| All routine visits and delivery | n/N (%) | n/N (%) | | | n/N (%) | | |
| 20 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 28 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| 36 weeks gestational age | n/N (%) | n/N (%) | | | n/N (%) | | |
| At the time of delivery | n/N (%) | n/N (%) | | | n/N (%) | | |
| Prevalence of molecular markers of DP resistance | n/N (%) | n/N (%) | | | n/N (%) | | |
| Prevalence of molecular markers of SP resistance | n/N (%) | n/N (%) | | | n/N (%) | | |
| Changes in measures of abundance | Mean Δ<br>(SD) | Mean ∆ | (SD) | p-<br>value | Mean Δ | (SD) | p-<br>value |
| Changes in vaginal/gut microbiome | xx (x.xx) | xx (x. | xx) | | xx (x.: | xx) | |
| Gestational weight gain per week (kg) <sup>c</sup> | xx (x.xx) | xx (x. | xx) | | xx (x.: | xx) | |

<sup>&</sup>lt;sup>a</sup> Reference group

<sup>&</sup>lt;sup>b</sup> Number of events (incidence per person year at risk)

<sup>&</sup>lt;sup>c</sup> Adjusted for baseline values

## 8 Safety and Tolerability Analyses (Objective 2)

Safety and tolerability will be evaluated during the period following the 1<sup>st</sup> dose of study drug administration through the end of the observation period (4 weeks post-partum) or premature study withdrawal.

## 8.1 Adverse Events

An adverse event will be defined as "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment" (ICH Guidelines E2A). An adverse event can further be broadly defined as any untoward deviation from baseline health, which includes:

- Worsening of conditions present at the onset of the study
- Deterioration due to the primary disease
- Intercurrent illness
- Events related or possibly related to concomitant medications

(International Centers for Tropical Disease Research Network Investigator Manual, Monitoring and Reporting Adverse Events, 2003).

At each scheduled and unscheduled visit to the clinic, study clinicians will assess patients according to a standardized case record form. A severity grading scale, based on toxicity grading scales developed by the NIH Divisions of AIDS (DAIDS) and the Division of Microbiology and Infectious Diseases (DMID) Pediatric Toxicity Tables, will be used to grade severity of all symptoms, physical exam findings, and laboratory results. All participants, regardless of treatment arm, will be assessed using the same standardized case record form. Adverse event monitoring will occur during the period when study drugs are given and up to 4 weeks following delivery. Data will be captured on the incidence of all adverse events, regardless of severity. For each adverse event identified as severity grade 3-4 or a serious adverse event (SAE), an additional adverse event report form will be completed.

#### 8.2 Serious Adverse Events

A Serious Adverse Event (SAE) will be defined as any adverse event that results in any of the following outcomes:

- Death
- Life-threatening adverse experience
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- Congenital malformation/birth defect
- Any other experience that suggests a significant hazard, contraindication, side effect or precaution that may require medical or surgical intervention to prevent one of the outcomes listed above
- Event that changes the risk/benefit ratio of the study

## 8.3 Analytical Methods

A modified intention-to-treat approach to all will be used, including all study participants who received at least one dose of study drugs, regardless of whether subsequently the intervention was not given for any reason. We will compare the proportions of study participants with vomiting following each dose of study drugs using generalized estimating equations with a log-binomial family and robust standard errors to account for repeated measures in the same study participant. We will compare the incidence of various adverse events using negative binomial regression models. The These models will include the logarithm of the follow-up time as an offset. We will translate the fitted coefficients and their confidence bounds into percentage effects with the formula 100\*[exp(coefficient)-1]. This approach is closely related to exponential survival models for analyzing events per follow-up time, but is better able to adjust for violated assumptions. Comparisons of incidence measures will be expressed at the incidence rate ratio (IRR) or the protective efficacy (PE = 1-IRR x 100%). A skeleton table for the presentation of safety and tolerability outcomes is presented in Table 11 below.

Table 11. Measures of safety and tolerability

| 0 | Treatment arm | | | | | | |
|---|---|---|---|---|---|---|---|
| Outcome | SP a | DP | | | SP+DP | | |
| Prevalence measures | Prevalence | Prevalence | RR<br>(95% CI) | p-<br>value | Prevalence | RR<br>(95% CI) | p-<br>value |
| Vomiting following administration of study drugs | | | | | | | |
| Observed after administration of 1st dose in clinic | n/N (%) | n/N (%) | | | | | |
| Reported after administration of 2 <sup>nd</sup> dose at home | n/N (%) | n/N (%) | | | | | |
| Reported after administration of 3rd dose at home | n/N (%) | n/N (%) | | | | | |
| Incidence measures | Events <sup>b</sup> | Events <sup>b</sup> | IRR<br>(95% CI) | p-<br>value | Events <sup>b</sup> | IRR<br>(95% CI) | p-<br>value |
| Individual adverse events of any severity c | | | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| Individual grade 3-4 adverse events <sup>c</sup> | | | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| XXXX | xx (x.xx) | xx (x.xx) | | | | | |
| All grade 3-4 adverse events | xx (x.xx) | xx (x.xx) | | | | | |
| Grade 3-4 adverse events possibly related to study drugs | xx (x.xx) | xx (x.xx) | | | | | |
| All serious adverse events | xx (x.xx) | xx (x.xx) | | | | | |

<sup>&</sup>lt;sup>a</sup> Reference group

<sup>&</sup>lt;sup>b</sup> Number of events (incidence per person year at risk)

<sup>&</sup>lt;sup>c</sup>Includes only those categories with at least five total events

## 9 References

- 1. Dellicour S, Tatem AJ, Guerra CA, Snow RW, ter Kuile FO. Quantifying the number of pregnancies at risk of malaria in 2007: a demographic study. PLoS Med 2010;7(1):e1000221. DOI: 10.1371/journal.pmed.1000221.
- 2. Desai M, ter Kuile FO, Nosten F, et al. Epidemiology and burden of malaria in pregnancy. Lancet Infect Dis 2007;7(2):93–104. (In eng). DOI: \$1473–3099(07)70021-X [pii]

## 10.1016/S1473-3099(07)70021-X.

- 3. Guyatt HL, Snow RW. Malaria in pregnancy as an indirect cause of infant mortality in sub-Saharan Africa. Trans R Soc Trop Med Hyg 2001;95(6):569-76. (https://www.ncbi.nlm.nih.gov/pubmed/11816423).
- 4. Walker PG, ter Kuile FO, Garske T, Menendez C, Ghani AC. Estimated risk of placental infection and low birthweight attributable to Plasmodium falciparum malaria in Africa in 2010: a modelling study. The Lancet Global health 2014;2(8):e460-7. DOI: 10.1016/S2214-109X(14)70256-6.
- 5. Gutman J, Kalilani L, Taylor S, et al. The A581G Mutation in the Gene Encoding Plasmodium falciparum Dihydropteroate Synthetase Reduces the Effectiveness of Sulfadoxine-Pyrimethamine Preventive Therapy in Malawian Pregnant Women. J Infect Dis 2015;211(12):1997-2005. DOI: 10.1093/infdis/jiu836.
- 6. Ranson H, N'Guessan R, Lines J, Moiroux N, Nkuni Z, Corbel V. Pyrethroid resistance in African anopheline mosquitoes: what are the implications for malaria control? Trends Parasitol 2011;27(2):91–8. DOI: 10.1016/j.pt.2010.08.004.
- 7. A head-to-head comparison of four artemisinin-based combinations for treating uncomplicated malaria in African children: a randomized trial. PLoS medicine 2011;8(11):e1001119. (Comparative Study

## **Multicenter Study**

#### Randomized Controlled Trial

Research Support, Non-U.S. Gov't) (In eng). DOI: 10.1371/journal.pmed.1001119.

- 8. White NJ. Intermittent presumptive treatment for malaria. PLoS Med 2005;2(1):e3. (In eng) (http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed &dopt=Citation&list\_uids=15696210).
- 9. Desai M, Gutman J, L'Lanziva A, et al. Intermittent screening and treatment or intermittent preventive treatment with dihydroartemisinin-piperaquine versus intermittent preventive treatment with sulfadoxine-pyrimethamine for the control of malaria during pregnancy in western Kenya: an open-label,

- three-group, randomised controlled superiority trial. Lancet 2015;386(10012):2507-19. DOI: 10.1016/S0140-6736(15)00310-4.
- 10. Kajubi R, Ochieng T, Kakuru A, et al. Monthly sulfadoxine-pyrimethamine versus dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria in pregnancy: A randomized controlled trial. The Lancet 2019.
- 11. Kakuru A, Jagannathan P, Muhindo MK, et al. Dihydroartemisinin-Piperaquine for the Prevention of Malaria in Pregnancy. N Engl J Med 2016;374(10):928–39. DOI: 10.1056/NEJMoa1509150.
- 12. Committee WHOMPA, Secretariat. Malaria Policy Advisory Committee to the WHO: conclusions and recommendations of eighth biannual meeting (September 2015). Malar J 2016;15:117. DOI: 10.1186/s12936-016-1169-x.
- 13. Chico RM, Moss WJ. Prevention of malaria in pregnancy: a fork in the road? Lancet 2015;386(10012):2454-6. DOI: 10.1016/S0140-6736(15)00325-6.
- 14. Chico RM, Chaponda EB, Ariti C, Chandramohan D. Sulfadoxine-Pyrimethamine Exhibits Dose-Response Protection Against Adverse Birth Outcomes Related to Malaria and Sexually Transmitted and Reproductive Tract Infections. Clin Infect Dis 2017;64(8):1043-1051. DOI: 10.1093/cid/cix026.
- 16. Schmiegelow C, Scheike T, Oesterholt M, et al. Development of a fetal weight chart using serial trans-abdominal ultrasound in an East African population: a longitudinal observational study. PLoS ONE 2012;7(9):e44773. DOI: 10.1371/journal.pone.0044773.
- 17. Villar J, Ismail LC, Victora CG, et al. International standards for newborn weight, length, and head circumference by gestational age and sex: the Newborn Cross-Sectional Study of the INTERGROWTH-21st Project. The Lancet 2014;384(9946):857-868.
- 18. Services DoANIoAaIDNIoHUDoHaH. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. (<a href="https://rsc.tech-res.com/docs/default-source/safety/daids\_ae\_grading\_table\_v2\_nov2014.pdf">https://rsc.tech-res.com/docs/default-source/safety/daids\_ae\_grading\_table\_v2\_nov2014.pdf</a>).